CLINICAL TRIAL: NCT05067920
Title: Correlation Between Cycle Threshold (Ct) Values in RT-PCR - SARS-CoV-2, Health Status and Laboratory Biomarkers in the Population of Medellin- Colombia Evaluated in a Specialized Laboratory
Brief Title: Correlation Between Cycle Threshold (Ct) Values in COVID-19, Health Status and Laboratory Biomarkers in the Population of Medellin- Colombia Evaluated in a Specialized Laboratory.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Antioquia (Other)
Collaborators: Laboratorio departamental de salud publica de Antioquia (Unknown); Sistema general de regalias (BPIN 2020000100152) (Unknown)
Responsible Party: Principal Investigator, Andres Felipe Zuluaga Salazar, Full profesor, senior researcher and head of the Department of Pharmacology and Toxicology in Antioquia University, Universidad de Antioquia
Other Study IDs: LIME01P2021
Record Dates: First submitted 2021-09-09; First posted 2021-10-05 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: Laboratory biomarkers; Health condition; CT value; COVID-19; Mitochondrial DNA
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic patients: 60 patients without COVID-19 symptoms related at the time of diagnosis.
  Interventions: Diagnostic Test: Levels of SARS-COV-2 antibodies; Diagnostic Test: rRT-PCR SARS-Cov-2; Diagnostic Test: Hematological and immunological biomarkers; Diagnostic Test: Mitochondrial DNA; Diagnostic Test: SARS-CoV-2 Viral Culturing; Diagnostic Test: Sequencing COVID-19
- Symptomatic patients: 60 patients with COVID-19 symptoms related at the time of diagnosis.
  Interventions: Diagnostic Test: Levels of SARS-COV-2 antibodies; Diagnostic Test: rRT-PCR SARS-Cov-2; Diagnostic Test: Hematological and immunological biomarkers; Diagnostic Test: Mitochondrial DNA; Diagnostic Test: SARS-CoV-2 Viral Culturing; Diagnostic Test: Sequencing COVID-19

INTERVENTIONS:
Diagnostic Test: Levels of SARS-COV-2 antibodies — Study of the SARS-COV-2 antibodies of COVID-19 IgM ( day 5th and 14th) and IgG ( day 14th and 28th)
Diagnostic Test: rRT-PCR SARS-Cov-2 — Real time RT-PCR for COVID-19 diagnosis at day 5th,14th and 28th
Diagnostic Test: Hematological and immunological biomarkers — Laboratory data measure at day 5th,14th and 28th: Hemogram, cytokine levels, ratio of CD4 + / CD8 + lymphocytes, and levels of dehydrogenase lactate, ferritin, D-dimer.
Diagnostic Test: Mitochondrial DNA — One time quantification mitochondrial DNA haplogroup.
Diagnostic Test: SARS-CoV-2 Viral Culturing — Probability of isolating SARS-Cov-2 in cell culture related to CT value above 32.
Diagnostic Test: Sequencing COVID-19 — Sequencing viral protein spike (S) COVID-19 related to CT value below 15.

SUMMARY:
This study will evaluate the correlation between the symptomaticity, Ct value, laboratory biomarkers associated to COVID-19 and the disease progression in hospitalized patients and outpatients with SARS-CoV2 infection diagnosed by RT-PCR assay for nasopharyngeal swab specimens in a specialized laboratory at Medellin,Colombia.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will undergo a serial of test related to COVID-19. Rh and blood type will be obtained using the Colombian ID card or official document.

All symptomatic and asymptomatic COVID19-positive patients will be evaluated for a period of 4 weeks at three different times of the study. In a single time, the mitochondrial DNA will be measured, and the variability in the CT value, hemogram, cytokine levels, ratio of CD4 + / CD8 + lymphocytes, levels of dehydrogenase lactate, ferritin and D-dimer, antibodies IgG and IgM, will be measured on day 5, day 14 and day 28. In addition, spike S protein sequencing and growing the virus in cell culture that meet specific criteria will be performed. A physician will do clinical follow up through the period of the study for each patient.

ELIGIBILITY:
Inclusion Criteria:

* People under 18 years old.
* Covid-19 diagnosis in the last seven days.
* Specimen analyzed at LIME laboratory
* Description of symptoms related to COVID-19

Exclusion Criteria:

* Immunocompromised patients
* Immunosuppressive treatments, chemotherapy or antiretroviral therapy
* Outpatient anticoagulation therapy
* Prior immunization for any vaccine in the last 3 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 confirmed patients with SARS-Cov-2 RT-PCR in Laboratorio Integrado de Medicina Especializada (LIME) or IPS Universitaria Clinica Leon XIII
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical immune response among COVID-19 patients related to CT value of rRT-PCR SARS-Cov-2 | Through study completion, an average of 4 months
  Calculated Ct value over 4 weeks, comparing the change in the immune status through the measurement of biomarkers

SECONDARY OUTCOMES:
Determine the duration of the positivity of the PCR test in asymptomatic and symptomatic patients through the follow-up | Through study completion, an average of 4 months
Evaluate differences in the titers of immunoglobulins M and G against anti-RBD domain of the protein S in SARS-CoV2 | Through study completion, an average of 4 months
Capacity of isolating the virus in cell culture with Ct> 32 by PCR in COVID-19 patients | Through study completion, an average of 4 months
Identification of polymorphic variants or mutations in COVID-19 patients | Through study completion, an average of 4 months
Mitochondrial DNA haplogroup relation in people infected with SARS CoV2 | Through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Andres F Zuluaga, MD, MSc, MeH, Principal Investigator — Universidad de Antioquia
Locations (1):
- Laboratorio Integrado de Medicina Especializada, Medellín, Antioquia, Colombia